CLINICAL TRIAL: NCT02313688
Title: The Relationship Between the Length of the Proximal Resection Margin and Long-term Survival for Adenocarcinomas of the Esophagogastric Junction (Siewert-II/Siewert-III)- Randomized Controlled Trial
Brief Title: Length of the Proximal Resection Margin for Siewert-II/Siewert-III Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Jian-Kun Hu, Prof. of Gastrointestinal Surgery Department., West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCH-GC-02
Record Dates: First submitted 2014-12-07; First posted 2014-12-10 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Stomach Neoplasms; Siewert Type II Adenocarcinoma of Esophagogastric Junction; Recurrence; Siewert Type III Adenocarcinoma of Esophagogastric Junction
Keywords: adenocarcinomas of esophagogastric junction; resection margin; length; prognosis
MeSH Terms: conditions — Stomach Neoplasms; Recurrence; Margins of Excision | interventions — Gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Group A: Patients in the Group A will underwent D2 total gastrectomy and with 3±0.5 cm lengthen proximal resection margin. Intraoperative frozen section will routinely performed to secure the tumor free resection margin.
  Interventions: Procedure: gastrectomy
- Group B (Experimental): Patients in the Group B will underwent D2 total gastrectomy and with 5±0.5 cm lengthen proximal resection margin. Intraoperative frozen section will routinely performed to secure the tumor free resection margin.
  Interventions: Procedure: gastrectomy

INTERVENTIONS:
Procedure: gastrectomy — Transabdominal (include transhiatal) D2 gastrectomy according JGCA gastric cancer treatment guidelines (2010, ver.3) and with 3±0.5 cm lengthen proximal resection margin.
  Arms: Group A
Procedure: gastrectomy — Transabdominal (include transhiatal) D2 gastrectomy according JGCA gastric cancer treatment guidelines (2010, ver.3) and with 5±0.5 cm lengthen proximal resection margin.
  Arms: Group B

SUMMARY:
The incidence of adenocarcinomas of the esophagogastric junction (AEJ) has increased rapidly during the past decades. By the Siewert classification, the AEJ is the tumor center located 5 cm above the anatomic cardia and 5 cm below it, which is divided into three individual subtypes. Complete tumor resection is the primary therapy strategies for tumors of the AEJ. The Japan Clinical Oncology Group 9502 (JCOG 9502) found that transabdominal or transhiatal approach gastrectomy has better survival outcomes compared with left thoracoabdominal approach surgery for Siewert II/III tumors. Transabdominal approach gastrectomy is recommended as the standard treatment strategy for Siewert II/III tumors by the guidelines of the Japanese Gastric Cancer Association (JGCA). However, the length of the proximal resection margin for Siewert-II/III tumors by transabdominal/transhiatal gastrectomy is still controversies. Previous study found that longer than 2cm proximal resection margin had better survival outcome than less than 2cm proximal resection margin for Siewert-II/III tumors. On the other sides, due to more advanced tumor stage of patients in China when compared with Japan and Korea. It is necessary to conduct a randomized control study to analyze the length of resection margin in advanced adenocarcinomas of esophagogastric junction.

Therefore, this study was aimed to include those Siewert II/III tumor patients in Gastrointestinal Surgery Department, West China Hospital, Sichuan University to analyze the relationship between the length of proximal resection margin and survival outcomes.

DETAILED DESCRIPTION:
Standard Operating Procedure (SOP)

1. Preoperative evaluation Patients satisfied with inclusion/exclusion criteria will be informed to join in the clinical study and signature the inform consent.
2. Randomization: Intraoperative evaluation found that transabdominal or transhiatal R0, D2 lymphadenectomy, total gastrectomy can be performed, the case will entrance into the Randomization period. Random numbers are computer-generated, with the third party applications.
3. Surgical procedures: The surgical treatments is adopted the total gastrectomy according to the Japanese Gastric Cancer treatments guidelines, 2010, Version 3. Patients in the Group A with 3cm length proximal resection margin and patients in the Group B with 5cm length proximal resection margin. Intraoperative frozen section will routinely performed to secure the tumor free resection margin. If the positive resection margin is found by the intraoperative frozen section, supplementary resection was depend on the characteristics of each patients. Whether these patients with supplementary resection, the length of supplementary resection and the times of the supplementary resection are all needed to record. The two study will take the similar surgical procedures except for the length of the resection margin.
4. Postoperative recovery: Postoperative recovery period need to collect those relevant parameters of all the patients. All the relevant parameters had definitely definition in the Case Report Form of this study which included the preoperative, intraoperative and postoperative clinicopathologic characteristics.
5. Follow-up: The follow-up of this study divide into two parts, the postoperative complications and survival outcomes. The postoperative complications is graded by the Clavien-Dindo classification. The survival outcomes included recurrence type, relapse free survival (months) and the overall survival (months).

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative endoscopy and biopsy confirmed upper third gastric adenocarcinoma (Siewert-II/Siewert-III), and predictively feasible of radical total gastrectomy;
2. Predictively resectable diseases, advanced gastric cancer, of preoperative staging JGCA 14th Edition cT2N0M0-T4aN3bM0, Ib-IIIc stage;
3. Age：≤75 years, or ≥18 years;
4. Without serious disease and malignance disease;
5. WHO performance score ≤2, ASA score ≤3;
6. No limit to sexual and race;
7. Informed consent required.

Exclusion Criteria:

1. Patients with other severe complications cannot tolerate surgery: such as severe heart and lung diseases, heart function below clinical stage 2, uncontrollable hypertension, pulmonary infection, moderate to severe COPD, chronic bronchitis, severe diabetes and / or renal insufficiency, severe hepatitis and / or function below the rank of CHILD B grade, and severe malnutrition, etc;
2. Patients treated with neoadjuvant chemotherapy or radiation therapy which might affect the efficacy observation;
3. Severity mental diseases;
4. Primary lesion cannot be resected in the pattern of transabdominal proximal gastrectomy, but for total gastrectomy, Whipple's procedure, or combined organ resection or with a transthoracic approach surgery;
5. After signature the Clinical trial agreement, patients and their agent will quit the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival | 3 years

SECONDARY OUTCOMES:
3-year overall survival | 3 years
Recurrence type | 3 years
The positive rate of proximal resection margin | Intraoperative
  Examined by the intraoperative frozen section

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Kun Hu, M.D. Ph.D., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China